CLINICAL TRIAL: NCT02503215
Title: Effects of Compression Stockings on Obstructive Sleep Apnea and Autonomic Nervous System in Patients Under Hemodialysis
Brief Title: Effects of Compression Stockings on Obstructive Sleep Apnea in Patients Under Hemodialysis
Acronym: EComStockOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Bruno Caldin da Silva, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21833413.0.0000.0068
Record Dates: First submitted 2014-12-26; First posted 2015-07-20 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Renal Failure Chronic Requiring Dialysis; Obstructive Sleep Apnea
Keywords: Hemodialysis; Obstructive sleep apnea; Compression stockings
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Stockings, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compression Stockings (Experimental): Patients will wear graduated lower limb compression stockings for a week. The investigators will evaluate if such procedure will cause better sleep performance
  Interventions: Device: Compression Stockings

INTERVENTIONS:
Device: Compression Stockings — To evaluate the effects of compression stockings on fluid shift and sleep apnea in hemodialysis patients with obstructive sleep apnea

SUMMARY:
To study the effects of compression stockings on sleep apnea in hemodialysis patients with diagnosed obstructive sleep apnea. The rationale of this study consists in the fluid shift theory, which consists in the nocturnal rostral fluid shift from legs, which causes upper airways edema.

The aim of this study is to evaluate if compression stockings could improve such nocturnal volume redistribution and, therefore, improve obstructive sleep apnea.

DETAILED DESCRIPTION:
Investigators will apply the following methods:

* Sleep study, performed through polysomnography
* Fluid redistribution, by bioimpedance analysis
* Autonomic nervous system evaluation, by spectral heart rate variability analysis.

The study protocol comprises two moments: baseline evaluation (in patients with diagnosed sleep apnea) and after using compression stockings for a one-week period.

ELIGIBILITY:
Inclusion Criteria:

* Patients under hemodialysis
* Patients with diagnosed obstructive sleep apnea

Exclusion Criteria:

* Congestive heart failure
* Urine output > 500 ml/day
* non-sinusal cardiac rhythm
* refusal to give written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno C Silva, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas 05302050, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Elias RM, Chan CT, Paul N, Motwani SS, Kasai T, Gabriel JM, Spiller N, Bradley TD. Relationship of pharyngeal water content and jugular volume with severity of obstructive sleep apnea in renal failure. Nephrol Dial Transplant. 2013 Apr;28(4):937-44. doi: 10.1093/ndt/gfs473. Epub 2012 Nov 7. PMID 23136217
- [Background] Kasai T, Motwani SS, Elias RM, Gabriel JM, Taranto Montemurro L, Yanagisawa N, Spiller N, Paul N, Bradley TD. Influence of rostral fluid shift on upper airway size and mucosal water content. J Clin Sleep Med. 2014 Oct 15;10(10):1069-74. doi: 10.5664/jcsm.4102. PMID 25317087
- [Background] White LH, Lyons OD, Yadollahi A, Ryan CM, Bradley TD. Effect of below-the-knee compression stockings on severity of obstructive sleep apnea. Sleep Med. 2015 Feb;16(2):258-64. doi: 10.1016/j.sleep.2014.12.005. Epub 2014 Dec 18. PMID 25620198
- [Background] Redolfi S, Arnulf I, Pottier M, Lajou J, Koskas I, Bradley TD, Similowski T. Attenuation of obstructive sleep apnea by compression stockings in subjects with venous insufficiency. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1062-6. doi: 10.1164/rccm.201102-0350OC. PMID 21836140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for sleep apnea from August to October 2014. Screening consisted of applying the Berlin Questionnaire. Patients at risk for sleep-disordered breathing were then submitted to polysomnography in order to confirm obstructive sleep apnea.
  Patients with apnea/hypopnea index > 5 were recruited.
Pre-assignment Details: Patients who did not have obstructive sleep apnea at the initial polysomnography evaluation were excluded from study. Additionally, patients who were unable to wear compression stockings or use positive airway pressure after enrollment were also excluded from study
Groups:
- Compression Stockings: Patients wore graduated lower limb compression stockings for a week. The investigators evaluated if such procedure caused better sleep performance
  Compression Stockings: To evaluate the effects of compression stockings on fluid shift and sleep apnea in hemodialysis patients with obstructive sleep apnea
Period: Overall Study
Arm/Group | Compression Stockings
Started | 17
Completed | 14
Not Completed | 3
Not completed — Unable to wear compression stockings | 1
Not completed — Unable to use positive airway pressure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Compression Stockings
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 14

OUTCOME MEASURES:

1. Primary Outcome: Change of Obstructive Apnea Severity Index Score From Baseline
Description: Apnea/Hypopnea index (AIH) was assessed by a validated polysomnography (EMBLA®S4500, Embla Systems Inc., Broomfield, CO, USA) at baseline and 1 week after compression stockings use. The observed results are expressed as median and interquartile range (25,75 percentiles):
  * AIH at baseline: 20.8 (14.2; 39.6) events/hour;
  * AIH after compression stockings use: 16.7 (3.5; 28.9) events/hour
Time Frame: 1 week
Population: Apnea/Hypopnea Index
Measure: Median (Inter-Quartile Range); unit: events/hour
Arm/Group | Compression Stockings
Number analyzed (Participants) | 14
events/hour
  Baseline | 20.8 [14.2 to 39.6]
  Compression Stockings | 16.7 [3.5 to 28.9]

2. Secondary Outcome: Change of Heart Rate Variability Change From Baseline
Description: Electrocardiogram performed during polysomnography examination will be downloaded to a specific software for heart rate variability assessment (Kubius HRV™, University of Eastern Finland, Finland), which provides spectral assessment of heart rate variability in its both components: low frequency (LF) and high frequency (HF). Patients who present higher LF/HF during the night compared to the beggining of the polysomnography exam have, by definition, increased sympathetic activity during the night. Such evaluation will be accessed in both baseline and after compression stockings use.
Time Frame: 1 week
Population: Overnight increase in LF/HF ratio at baseline: 11/12 patients (92%) Overnight increase in LF/HF ratio after compression stockings use: 7/12 patients (58%)
Measure: Number; unit: percentage of participants
Arm/Group | Compression Stockings
Number analyzed (Participants) | 12
percentage of participants
  Baseline | 92
  Compression Stockings | 58

3. Secondary Outcome: Change in Fluid Distribution From Baseline
Description: Segmental and total body water will be non-invasively assessed before sleeping and after awakening by a bioimpedance device (InBody S10 Analyser™, Biospace, South Korea), which will provide information regarding nighttime fluid shift at baseline and after compression stocking use. The amount of water, expressed in liters, is assessed in both extra and intracellular components.
Time Frame: 1 week
Population: Volume distribution evaluated by bioimpedance analysis evaluated fluid shift from the legs at baseline and after wearing compression stockings. The amount overnight fluid that moved rostrally from the legs is depicted below (results expressed as mean ± standard deviation):
  * Baseline: 571.4 ± 389.6 ml
  * Compression stockings: 517.9 ± 452.2 ml
Measure: Mean (Standard Deviation); unit: mililiters
Arm/Group | Compression Stockings
Number analyzed (Participants) | 14
mililiters
  Baseline | 571.4 (389.6)
  Compression Stockings | 517.9 (452.2)

ADVERSE EVENTS:
Time Frame: Data regarding adverse events were collected during the one-week period while patients wore the compression stockings. Events assessed: dyspnea, and lower limbs pain.
Arm/Group | Compression Stockings
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
During heart rate variability analysis, two patients had techinical problems during electrocardiogram aquisition and could not habe their data analysed and were therefore excluded from final results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No